CLINICAL TRIAL: NCT01108055
Title: A Phase II Study of Pazopanib in Combination With Weekly Paclitaxel in Refractory Urothelial Cancer
Brief Title: Phase II Pazopanib in Combination With Weekly Paclitaxel in Refractory Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sandy Srinivas (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Sandy Srinivas, Associate Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-17472; SU-04152010-5683 (Other: Stanford University); BLDR0010 (Other: OnCore)
Record Dates: First submitted 2010-04-15; First posted 2010-04-21 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Bladder Cancer; Bladder (Urothelial, Transitional Cell) Cancer; Bladder (Urothelial, Transitional Cell) Cancer Superficial (Non-Invasive); Bladder (Urothelial, Transitional Cell) Cancer Resectable (Pre-Cystectomy); Bladder (Urothelial, Transitional Cell) Cancer Metastatic or Unresectable
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — pazopanib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pazopanib + paclitaxel (Experimental): Cycle of 28 days. Pazopanib: 800mg daily
  Cycle of 28 days Paclitaxel: 80mg/m2 on days 1,8 and 15
  Interventions: Drug: Pazopanib (GW786034); Drug: Paclitaxel

INTERVENTIONS:
Drug: Pazopanib (GW786034) — Cycle of 28 days. Pazopanib: 800mg/day
  Other Names: GW786034
Drug: Paclitaxel — Cycle of 28 days Paclitaxel: 80mg/m2 days 1,8 and 15
  Other Names: Taxol

SUMMARY:
We will combine an oral investigational vascular endothelial growth factor (VEGF inhibitor) called pazopanib which is being studied in kidney cancer will be combined with standard chemotherapy called taxol in patients with relapsed recurrent urothelial cancer.

DETAILED DESCRIPTION:
Based on the results from the Phase 1 study of pazopanib combined with paclitaxel and the activity of paclitaxel in urothelial cancer, testing this regimen in a disease where there is an unmet need appears appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed transitional cell carcinoma (TCC) of the urothelium (bladder, renal pelvis, ureter, or urethra). Mixed histology is allowed as long as the predominant histology is TCC
2. First recurrence after treatment with a maximum of two chemotherapeutic regimens.
3. Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow up.

   Procedures conducted as part of the subject's routine clinical management (eg, blood count, imaging study) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol.
4. Age ≥ 18 years
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
6. Measurable disease criteria by RECIST criteria
7. Adequate organ system function as defined below

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
   2. Hemoglobin ≥ 9 g/dL
   3. Platelets ≥ 100 X 10^9/L
   4. Prothrombin time (PT) or international normalized ratio (INR) ≤ 1.2 x upper limit of normal (ULN)
   5. Total bilirubin ≤ 1.5 x ULN
   6. aspartate aminotransferase (AST) and Alanine Aminotransferase (ALT)≤ 2.5 x ULN
   7. Serum creatinine ≤ 1.8 mg/dL
   8. Urine Protein to Creatinine Ratio (UPC) < 1
8. A female is eligible to enter and participate in this study if she is of non-childbearing potential (ie, physiologically incapable of becoming pregnant). This includes any female who has had:

   * A hysterectomy
   * A bilateral oophorectomy (ovariectomy)
   * A bilateral tubal ligation
   * Menopause

Childbearing potential females must have a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agree to use adequate contraception. Adequate acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow:

* An intrauterine device with a documented failure rate of less than 1% per year.
* Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
* Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product.
* Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide).

Exclusion Criteria:

1. History of other malignancies within 5 years prior to Day 1 except for tumors with a negligible risk for metastasis or death, such as adequately controlled basal cell carcinoma, squamous-cell carcinoma of the skin, carcinoma in situ of the cervix, early-stage bladder cancer, or low-grade endometrial cancer Malignancies that have undergone a putative surgical cure (ie, localized prostate cancer post-prostatectomy) within 5 years prior to Day 1 may be discussed with the Medical Monitor
2. History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug.
3. Clinically significant gastrointestinal abnormalities that may increase the risk for GI bleeding
4. Clinically significant gastrointestinal abnormalities that may affect absorption of the investigational product
5. Presence of uncontrolled infection.
6. Prolongation of corrected QT interval (QTc) > 480 milliseconds. On antiarrhythmics or medications known to prolong QT interval
7. History of any one or more of the following cardiovascular conditions within the past 6 months:

   * Cardiac angioplasty or stenting
   * Myocardial infarction
   * Unstable angina
   * Coronary artery by-pass graft surgery
   * Symptomatic peripheral vascular disease
   * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
8. Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥ 140 mmHg or diastolic blood pressure (DBP) of ≥ 90mm Hg].
9. History of cerebrovascular accident, hemoptysis, cerebral hemorrhage, clinically significant GI bleed, pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months
10. Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture
11. Evidence of active bleeding or bleeding diathesis.
12. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to procedures.
13. Patients on strong CYP3A4 inhibitors
14. Uncorrected abnormal electrolytes: K, Mg and Ca
15. Prior treatment with taxane chemotherapy
16. Treatment with any of the following anti-cancer therapies:

    * radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR
    * chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-04; Primary Completion 2015-01 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sandy Srinivas, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - Karmanos Cancer Institute, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pazopanib + Paclitaxel: A trial combining paclitaxel with pazopanib, a commonly used anti-angiogenic agent with significant anti-tumor activity in various solid tumors.
Period: Overall Study
Arm/Group | Pazopanib + Paclitaxel
Started | 43
Eligible and Started Treatment | 32
Completed | 28
Not Completed | 15
Not completed — Ineligible | 11
Not completed — Not evaluable- didn't complete treatment | 4

BASELINE CHARACTERISTICS:
Arm/Group | Pazopanib + Paclitaxel
Number analyzed (Participants) | 32
Age, Continuous [Mean (Full Range); unit: years] | 67 [29 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 23
  More than one race | 0
  Unknown or Not Reported | 2
Prior Treatment Cycles [Median (Full Range); unit: Cycles] — A full treatment cycle is defined as 28 days.
  Cycles | 4 [1 to 14]
Sites of Primary Tumor [Count of Participants; unit: Participants]
  Bladder | 15
  Renal Pelvis | 11
  Ureter | 6
Number of prior chemotherapies [Count of Participants; unit: Participants]
  1 | 13
  2 | 19
Time from last chemotherapy [Count of Participants; unit: Participants]
  < 3 months | 15
  > 3 months | 17
Bellmunt Score [Count of Participants; unit: Participants]
  0 | 7
  1 | 14
  2 | 11
  3 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response
Description: The tumor response rate was assessed per the Response Evaluation Criteria In Solid Tumors (RECIST). RECIST criteria are a set of published rules that define when cancer patients improve ("respond"); stay the same ("stable"); or worsen ("progression") during treatments. RECIST criteria offer a simplified and conservative extraction of imaging data suitable for wide application in clinical trials. The criteria presume that linear measures are an adequate substitute for 2-dimensional (2D) methods and includes 4 response categories:
  * Complete response (CR) = Disappearance of all target lesions
  * Partial response (PR) = 30% decrease in the sum of the longest diameter of target lesions
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions
  * Stable disease (SD) = Small changes that do not meet above criteria Objective tumor response means those with response better than stable disease, ie, complete response (CR) + partial response (PR).
Time Frame: Every 8 weeks
Population: The outcome is reported as subjects with CR (complete response) + PR (partial response).
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib + Paclitaxel
Number analyzed (Participants) | 32
Participants | 15

2. Secondary Outcome: Progression-free Survival (PFS)
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pazopanib + Paclitaxel
Number analyzed (Participants) | 32
Months | 6.2 [5.6 to 7.6]

3. Secondary Outcome: Overall Response Rate
Description: The tumor response rate was assessed per the Response Evaluation Criteria In Solid Tumors (RECIST). RECIST criteria are a set of published rules that define when cancer patients improve ("respond"); stay the same ("stable"); or worsen ("progression") during treatments. RECIST criteria offer a simplified and conservative extraction of imaging data suitable for wide application in clinical trials. The criteria presume that linear measures are an adequate substitute for 2-dimensional (2D) methods and includes 4 response categories:
  * Complete response (CR) = Disappearance of all target lesions
  * Partial response (PR) = 30% decrease in the sum of the longest diameter of target lesions
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions
  * Stable disease (SD) = Small changes that do not meet above criteria Tumor response rate by each response criteria.
Time Frame: 4 years
Population: Does not include participants who did not complete 2 cycles of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib + Paclitaxel
Number analyzed (Participants) | 28
Participants
  Complete Response (CR) | 3
  Partial Response (PR) | 12
  Stable Disease (SD) | 11
  Progressive Disease (PD) | 2

4. Secondary Outcome: Overall Survival
Description: Overall survival is reported as the median survival of the evaluable subjects (ie, completed 2 cycles of treatment).
Time Frame: 4 years
Population: Does not include participants who did not complete 2 cycles of treatment.
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Pazopanib + Paclitaxel
Number analyzed (Participants) | 28
Months | 10 [5.7 to 16]

5. Secondary Outcome: Median Overall Survival (OS) by Bellmunt Score
Description: Comparison between the participant's baseline Bellmunt prognostic risk factor score and survival rates.
  The Bellmunt prognostic risk factor score is a tool that is often used to predict treatment outcomes before initiating a secondline treatment regimen.
  The risk factors used to calculate the Bellmunt score include:
  * Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1
  * Presence of liver metastases
  * Presence of visceral involvement (defined as liver, lung, bone or any non-lymph node)
  * Lymph node-only involvement
  * Hemoglobin concentration < 10 g/dL
  The score is calculated based on the presence of 0; 1; 2; or 3 of the above prognostic factors. This outcome reports median overall survival based on whether the participant had 0; 1; 2; or 3 prognostic factors.
Time Frame: 4 years
Population: Include all 32 participants, regardless of completing 2 cycles of treatment.
Measure: Median (Full Range); unit: Months
Arm/Group | Pazopanib + Paclitaxel
Number analyzed (Participants) | 32
Months
  Bellmunt Score of 0: number analyzed (Participants) | 7
  Bellmunt Score of 0 | 13.8 [6 to 24]
  Bellmunt Score of 1: number analyzed (Participants) | 14
  Bellmunt Score of 1 | 8 [2 to 55]
  Bellmunt Score of 2: number analyzed (Participants) | 11
  Bellmunt Score of 2 | 7.7 [1 to 21]
  Bellmunt Score of 3: number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Pazopanib + Paclitaxel
Serious Adverse Events (participants affected / at risk) | 15/32
Other Adverse Events (participants affected / at risk) | 20/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pazopanib + Paclitaxel (N=32)
electrolyte imbalance (Investigations) | 1 (1)
wound complication, non infectious (Skin and subcutaneous tissue disorders) | 1 (1)
gastrointestinal fistula (Gastrointestinal disorders) | 1 (1)
febrile neutropenia (Infections and infestations) | 2 (2)
infection with grade 3 or 4 neutrophils (Infections and infestations) | 2 (2)
Fever (General disorders) | 2 (2)
bacterial pneumonia (Infections and infestations) | 1 (1)
infection with normal ANC (Infections and infestations) | 1 (1)
Cord compression (Musculoskeletal and connective tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pazopanib + Paclitaxel (N=32)
Fatigue (General disorders) | 15 (35)
Weight loss (Metabolism and nutrition disorders) | 4 (5)
Insomnia (General disorders) | 2 (2)
diaphoresis (Skin and subcutaneous tissue disorders) | 2 (2)
fever (Infections and infestations) | 1 (1)
anorexia (Gastrointestinal disorders) | 8 (9)
diarrhea (Gastrointestinal disorders) | 5 (8)
nausea (Gastrointestinal disorders) | 4 (6)
Vomiting (Gastrointestinal disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 3 (3)
dysgeusia (Gastrointestinal disorders) | 3 (4)
Distension/bloating, abdominal (Gastrointestinal disorders) | 2 (2)
Mucositis/stomatitis - oral cavity (Gastrointestinal disorders) | 2 (2)
salivary gland changes/saliva (Gastrointestinal disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 1 (1)
GI, other (Gastrointestinal disorders) | 1 (1)
lukocytes (Blood and lymphatic system disorders) | 9 (12)
Platelets (Blood and lymphatic system disorders) | 8 (16)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 4 (8)
anemia (Blood and lymphatic system disorders) | 6 (16)
lymphopenia (Blood and lymphatic system disorders) | 6 (27)
hemolysis (Blood and lymphatic system disorders) | 2 (2)
pain, back (General disorders) | 6 (7)
Pain, abdomen NOS (General disorders) | 5 (7)
Pain, head/headache (General disorders) | 4 (4)
Pain, chest/thorax NOS (General disorders) | 3 (3)
Pain Extremity-limb (General disorders) | 2 (2)
Pain, chest wall (General disorders) | 1 (1)
Pain, oral cavity (General disorders) | 1 (1)
Creatinine, increased (Investigations) | 7 (13)
Alt, SGPT (Investigations) | 6 (8)
hyperglycemia (Investigations) | 6 (9)
hypoalbuminemia (Investigations) | 5 (7)
hypocalcemia (Investigations) | 4 (8)
hypokalemia (Investigations) | 4 (7)
alkaline phosphatase (Investigations) | 3 (4)
hypomagnesemia (Investigations) | 3 (3)
hyponatremia (Investigations) | 3 (5)
hyperbilirubinemia (Investigations) | 2 (2)
hyperkalemia (Investigations) | 2 (4)
proteinuria (Investigations) | 2 (2)
Bicarbonate, serum-low (Investigations) | 1 (1)
Glomerular Filtration rate (Investigations) | 1 (4)
hypophosphatemia (Investigations) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 7 (9)
Dizziness (Nervous system disorders) | 5 (5)
Cognitive distrubance (Nervous system disorders) | 1 (1)
memory impariment (Nervous system disorders) | 1 (1)
Mood alteration - Anxeity (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (10)
pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hair loss/alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (4)
bruising (in absence of grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1 (2)
Nail Changes (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Infection with unknown ANC - Bladder (Infections and infestations) | 1 (1)
Infection with unknown ANC - Sinus (Infections and infestations) | 1 (1)
infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 1 (1)
hemorrhage/bleeding (General disorders) | 2 (5)
hemorrhage, GI - Varices (Gastrointestinal disorders) | 1 (1)
hemorrhage, GU - bladder (Renal and urinary disorders) | 1 (1)
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Musculoskeletal/Soft Tissue - other (Musculoskeletal and connective tissue disorders) | 2 (2)
muscle weakness, extraocular (Musculoskeletal and connective tissue disorders) | 1 (1)
muscle weakness, whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 3 (4)
vascular - other (Vascular disorders) | 1 (1)
hypertension (Cardiac disorders) | 3 (3)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Edema: head and neck (Blood and lymphatic system disorders) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 1 (1)
growth and development- other (General disorders) | 1 (1)
vision-flashing lights/floaters (Eye disorders) | 1 (1)
gynecomastia (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No